CLINICAL TRIAL: NCT06538415
Title: To Determine Whether Adding Polyphenol-rich Pulses to Daily Diet Improves Skin Health by Reshaping the Skin Microbiome and Lipids, and Reducing Oxidative Stress and Inflammation in Women
Brief Title: Adding Polyphenol-rich Pulses to Daily Diet Improves Skin Health by Reshaping the Skin Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB202401105
Record Dates: First submitted 2024-07-26; First posted 2024-08-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Pulse; Women; Skin health

STUDY DESIGN:
Intervention Model Description: This trial will use a randomized, controlled, parallel design. Control type I error α = 0.05 (two-tailed) and type II error β =0.2. Assume an equal number of participants in the two groups. The calculated sample size is 20 per group. Factoring in a 20% dropout rate, 50 women will be enrolled in this study using a parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse Diet (Experimental): Participants will consume cooked pulse (112 calories -lentils, red kidney beans, black beans, and pinto beans) during 14 weeks.
  Interventions: Other: Pulse Diet
- Control Rice Diet (Active Comparator): Participants will consume cooked rice (112 calories) during 14 weeks.
  Interventions: Other: Control Rice Diet

INTERVENTIONS:
Other: Pulse Diet — Participants will consume cooked pulse (112 calories -lentils, red kidney beans, black beans, and pinto beans) during 14 weeks.
  Arms: Pulse Diet
Other: Control Rice Diet — Participants will consume cooked rice (112 calories) during 14 weeks.
  Arms: Control Rice Diet

SUMMARY:
Skin health is influenced by the microbiome, lipids, oxidative stress, inflammation, and UV exposure. A 14-week trial with 50 women aged 45-65 will test if polyphenol-rich pulses improve skin health by affecting these factors. Using a white rice control diet, the study will measure skin parameters and analyze correlations with changes in lipids and microbiome, potentially proving the benefits of pulses.

DETAILED DESCRIPTION:
Human skin is the largest organ in the body. The slow deterioration of skin appearance and its barrier function are the most prominent signs of human ageing. Cutaneous factors (microbiome and lipids) have immediate and direct impacts on skin health and functions. Intrinsic factors (oxidative stress and inflammation) and extrinsic ones (mostly UV irritation due to sun exposure) affect the skin chronically. Our preliminary research showed that six weeks of cranberry juice intake improved part of women's skin health parameters and decreased oxidative stress. Its activities on the skin correlated with changes in skin microbiome and epidermal lipids. Pulses, especially lentils and beans, are rich sources of polyphenols and fibers. However, there is no clinical evidence on whether adding a serving of cooked mixed pulses with high polyphenol content (lentils, red kidney bean, black beans, and pinto beans) to the diet affects skin health and the underlying causes of skin aging. Women make over 90% of the decisions on food purchases for their families. Skin health is a major concern for women because skin aging becomes visibly noticeable after age 30. The investigators hypothesize that polyphenol-rich pulses improve skin health by reshaping the cutaneous microbiome and lipids and suppressing inflammation and oxidative stress. This hypothesis will be tested in a 14-week clinical trial in 50 women aged 45-65 using a randomized controlled parallel design. The control diet will be formulated using white rice to match the calories and macronutrients of mixed pulses.

ELIGIBILITY:
Inclusion Criteria:

* BMI (18.5-29.9)
* Body weight ≥110 pounds
* Fitzpatrick skin type 2 and 3.

Exclusion Criteria:

* pregnancy
* breast-feeding
* impaired fasting glucose
* frequent alcohol use
* history of skin cancer
* sunbathing and the use of tanning bed, intake of vitamin/mineral supplements
* habitual high intake of fruits (≥ 2 cups daily)
* intake of medication that might influence the outcome of the study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin sensitivity after UV radiation | 100 days
  Irradiation will be applied to dorsal skin (back, scapular region not typically exposed to the sun) with 2 times of minimal erythema dose using an FDA approved UVB phototherapy light and a UV light meter. At baseline, after 56 and 112 days, skin color will be measured before and 24 hours after irradiation. Skin color will be evaluated by a colorimeter. The a*-value (red/green-axis) is a measure of reddening (erythema).

SECONDARY OUTCOMES:
skin transepidermal water loss | 100 days
  Skin transepidermal water loss will be measured using a Tewameter to evaluate the water barrier function of the skin. The Tewameter measures the density gradient of the water evaporation from the skin (g/h/m^2).
skin erythema and melanin index | 100 days
  Skin erythema and melanin index ((Arbitrary Mexameter Units on a scale of 0-999) will be assessed with Mexameter. These two components are mainly responsible for the color of the skin. They are measured by reflectance.
inflammation biomarkers | 100 days
  * Plasma concentration levels (pg/mL) of IL-6 proteins will be analyzed as inflammation biomarkers using ELISA kits.
  * Plasma concentration levels (mg/mL) of C-reactive proteins will be analyzed as inflammation biomarkers using ELISA kits.
oxidative stress biomarkers | 100 days
  Concentration of Malondialdehyde (nmol/mL) in plasma will be determined as a marker of lipid peroxidation using a photometric method.
skin microbiome | 100 days
  For skin swabbing, a 3x3-cm square on a forearm will be swabbed with a cotton swab soaked in 0.9% sodium chloride with 0.1% Tween-20 in a Z-stroke manner
skin hydration | 100 days
  Skin hydration (Arbitrary Units (AU) on a scale of 0-120) will be measured using a Skin Corneometer.
skin pH | 100 days
  Skin pH will be measured using a Skin-pH-Meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Food Science and Human Nutrition, Gainesville, Florida, United States